CLINICAL TRIAL: NCT04843137
Title: Investigating the Acute Effects of Transcutaneous Electrical Stimulation Parameters on Neural Circuits, Motoneuron Behavior and Motor Performance in Individuals With Cervical Spinal Cord Injury
Brief Title: Acute Mechanisms of Cervical Transcutaneous Electrical Stimulation of the Spinal Cord
Status: Withdrawn | Type: Observational
Why Stopped: Closed study at UofL, may reopen at new institution in the future. No participants have enrolled
Sponsor: University of Louisville (Other)
Responsible Party: Sponsor
Other Study IDs: 20.0593
Record Dates: First submitted 2021-04-06; First posted 2021-04-13 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Individuals with cervical spinal cord injury: Cohort of individuals who have experiences a chronic spinal cord injury at the cervical level (specifically C5-C7).
  Interventions: Device: Cervical Transcutaneous Electrical Spinal Cord Stimulation

INTERVENTIONS:
Device: Cervical Transcutaneous Electrical Spinal Cord Stimulation — Surface electrodes are placed over the cervical spinal cord. Constant current is delivery through these electrodes. Stimulation frequency and electrode configuration are manipulated, and outcome measures are recorded.
  Other Names: tcES

SUMMARY:
The purpose of this study is to examine how delivery of subthreshold electrical stimulation of the spinal cord alters the excitability of neural pathways and consequently movement performance in healthy and spinal cord injured individuals. Specifically, we assess how stimulation parameters such as electrode configurations and stimulation frequency affect spinal excitability, corticospinal excitability, intracortical excitability, motor unit properties and force production. This study is not an intervention study, but a mechanistic study trying to shed light on how this novel neuromodulatory technique acutely affects the central nervous system.

ELIGIBILITY:
Inclusion Criteria:

* cervical level injury (C5 to C7)
* at least 1 year post-injury

Exclusion Criteria:

* individuals with damage to the nervous system other than to the spinal cord
* pregnant women (effects of stimulation on the fetus are unknown).

Transcranial magnetic stimulation-specific exclusion criteria:

* participants with active or inactive implants including cardiac pacemakers, implantable defibrillators, ocular implants, deep brain stimulators, vagus nerve stimulator, and implanted medication pumps
* participants with conductive, ferromagnetic or other magnetic-sensitive metals implanted in their head
* participants with a history of seizures or epilepsy
* participants taking any medication which may reduce seizure threshold

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with chronic, cervical spinal cord injury.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-02-22 (Actual)

PRIMARY OUTCOMES:
Motor evoked potentials recruitment curves | Assessment up to 4 hours each visit; up to 4 visits per individual (32 hours)
  Motor evoked potentials are obtained to assess changes in the input/output properties of the corticospinal tract during delivery of tcES. Comparisons are made between no stimulation and stimulation at different frequencies, or with different electrode configurations. This assessment is repeated for different muscles on different days.
Intracortical excitability | Assessment up to 4 hours each visit; up to 4 visits per individual (32 hours)
  Paired stimulation of the motor cortex is used to assess short interval intracortical inhibition intracortical facilitation during delivery of tcES. Comparisons are made between no stimulation and stimulation at different frequencies, or with different electrode configurations. This assessment is repeated for different muscles on different days.
Intramuscular coherence | Assessment up to 4 hours each visit; up to 4 visits per individual (32 hours)
  High-density surface electromyography is used to decompose motor units and assess changes in intramuscular coherence during performance of a motor task in the presence of tcES. Comparisons are made between no stimulation and stimulation at different frequencies, or with different electrode configurations. This assessment is repeated for different muscles on different days.
Force control | Assessment up to 4 hours each visit; up to 4 visits per individual (32 hours)
  Force control during a variety of motor tasks is assessed during delivery of tcES. Comparisons are made between no stimulation and stimulation at different frequencies, or with different electrode configurations within each session. This assessment is repeated for different muscles on different days.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica D'Amico, PhD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Kentucky Spinal Cord Injury Research Centre, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No